CLINICAL TRIAL: NCT00967863
Title: Phase III Study Comparing Irradiation at a Dose of 80 Gy to Irradiation at 70 Gy in Unfavorable Prostate Cancers Associated With Prolonged Hormonal Therapy
Brief Title: Radiation Therapy in Treating Patients Receiving Hormone Therapy for Prostate Cancer (GETUG-AFU 18)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000649028 UC-0160/0706; FRE-FNCLCC-GETUG-18/0706; 2008-A00529-46 (Other: ANSM); EU-20966
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients undergo 80 Gy of conformal or intensity-modulated radiotherapy 5 times a week for 7-8 weeks.
  Interventions: Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy
- Arm II (Experimental): Patients undergo 70 Gy of conformal or intensity-modulated radiotherapy 5 times a week for 7-8 weeks.
  Interventions: Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Radiation: 3-dimensional conformal radiation therapy — Patients undergo radiotherapy
Radiation: intensity-modulated radiation therapy — Patients undergo radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. It is not yet known which dose of radiation therapy is more effective in treating patients with prostate cancer.

PURPOSE: This randomized phase III trial is comparing two radiation therapy regimens in treating patients with prostate cancer receiving hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the impact of increasing the radiation dose 10 Gy on biochemical or clinical progression-free survival at 5 years in patients with unfavorable-risk prostate cancer receiving prolonged hormone therapy.

Secondary

* Evaluate overall and specific survival.
* Assess acute and late toxicities of different modalities (conformal or intensity-modulated radiotherapy).
* Evaluate toxicities of the different doses with respect to hormonal therapy.
* Assess the quality of life (QLQ-C30 and PR 25).

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo 80 Gy of conformal or intensity-modulated radiotherapy 5 times a week for 7-8 weeks.
* Arm II: Patients undergo 70 Gy of conformal or intensity-modulated radiotherapy 5 times a week for 7-8 weeks.

In both arms, patients receive goserelin subcutaneously once every 3 months for up to 3 years.

After completion of study treatment, patients are followed up periodically for 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Unfavorable disease, defined by at least 1 of the following criteria:

    * Clinical stage T3 or T4
    * Gleason score ≥8
    * Serum prostate-specific antigen (PSA) ≥20 ng/mL and ≤100 ng/mL
* pN0 disease allowed if lymphadenectomy performed before patient began hormone therapy
* No pelvic lymph nodes ≥15 mm by CT scan or MRI
* No axillary lymph node involvement (pN1)
* No bone metastasis
* Must be starting hormonal treatment on or up to 6 months before beginning radiotherapy

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy >5 years
* Must be enrolled in a social security program
* No other cancer, except basal cell skin cancer, that has been treated or relapsed within the past 5 years
* No severe uncontrolled hypertension (systolic BP ≥160 mm Hg or diastolic BP ≥90 mm Hg)
* No contraindication to luteinizing hormone-releasing hormone agonists
* No contraindication to pelvic irradiation (e.g., scleroderma, chronic inflammatory gastrointestinal disease)
* No hip prosthesis
* Must not be deprived of liberty or under guardianship
* No geographical, social, or psychological reasons that would preclude follow up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior pelvic irradiation
* At least 3-4 months since prior transurethral resection
* No other prior surgery for prostate cancer
* No concurrent participation in another clinical trial which would require approval upon entry to this trial

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-10 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Biochemical or clinical progression-free survival at 5 years | 5 years

SECONDARY OUTCOMES:
Overall and specific survival | 10 years
Acute and late toxicity | 10 years
Quality of life as measured by QLQ-C30 and PR 25 questionnaires | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Christophe HENNEQUIN, PhD, Principal Investigator — Hopital Saint-Louis
Locations (25):
- France (25):
  - Institut de Cancérologie de l'Ouest Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre hospitalier Métropole Savoie, Chambéry
  - Clinique Léonard de Vinci, Chambray-lès-Tours
  - CHU Henri Mondor, Créteil
  - Centre Léon Bérard, Lyon
  - Hopital La Timone, Marseille
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Centre Val D'Aurelle, Montpellier
  - Centre Azureen de Cancerologie, Mougins
  - Chr Orleans, Orléans
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO - HPCA, Plérin
  - Hôpital Jean Bernard - CHU de Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Gauducheau, Saint-Herblain
  - Hia Begin, Saint-Mandé
  - Institut de Cancérologie LUCIEN NEUWIRTH, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Clinique PASTEUR, Toulouse
  - Ch Bretonneau, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Kim S, Kong JH, Lee Y, Lee JY, Kang TW, Kong TH, Kim MH, You SH. Dose-escalated radiotherapy for clinically localized and locally advanced prostate cancer. Cochrane Database Syst Rev. 2023 Mar 8;3(3):CD012817. doi: 10.1002/14651858.CD012817.pub2. PMID 36884035
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00967863